CLINICAL TRIAL: NCT02378740
Title: A Prospective, Block Randomized, Double-Blind Placebo-Controlled Trial of Ketamine in Patients Undergoing Anterior Cervical Discectomy and Fusion
Brief Title: Ketamine in Patients Undergoing Anterior Cervical Discectomy and Fusion
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI has left the University
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00102734
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Anesthesia; Pain; Surgery
Keywords: Anesthesia; Cervical Fusion; Quality of Recovery; Ketamine Infusion
MeSH Terms: conditions — Pain; Klippel-Feil Syndrome | interventions — Sodium Chloride; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (.9 sterile normal saline) administered IV
  Interventions: Drug: Saline
- Ketamine (Active Comparator): The study drug (either ketamine or saline) will be administered from the beginning of anesthesia through the commencement of wound closure to provide the following dose of ketamine:
  0.5 mg/kg loading dose 8.3 mcg/kg/min (0.5 mg/kg/hr) infusion
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Saline — The study drug (either ketamine or saline) will be administered from the beginning of anesthesia through the commencement of wound closure to provide the following dose of ketamine:
  0.5 mg/kg loading dose 8.3 mcg/kg/min (0.5 mg/kg/hr) infusion
  Arms: Placebo
Drug: Ketamine — The study drug (either ketamine or saline) will be administered from the beginning of anesthesia through the commencement of wound closure to provide the following dose of ketamine:
  0.5 mg/kg loading dose 8.3 mcg/kg/min (0.5 mg/kg/hr) infusion
  Arms: Ketamine

SUMMARY:
Ketamine is an IV anesthetic with non-opioid analgesic properties that has been shown to reduce pain while also decreasing intraoperative and postoperative opioid requirements when used in subanesthetic doses after a variety of surgical procedures.1 It is a non-competitive antagonist of N-methyl-D-aspartate (NMDA) receptors, and by this mechanism ketamine is believed to block the development of central sensitization and wind-up phenomenon,2,3 which may be helpful in preventing acute and chronic pain after repetitive insults. In a systematic review of ketamine as an adjuvant to opioid analgesia, low-dose ketamine was found to be a useful addition to standard postoperative pain management practice with opioids in 54% of studies.1 The studies that did not show a significant effect were in patient populations with low opioid requirements. Therefore, it has been suggested that future clinical trials be focused on patient populations with significant post-operative pain, such as spine surgery and major orthopedic surgery not amenable to regional analgesia, and postoperative pain in patients on chronic preoperative opioid therapy.1

There are few studies examining outcomes after ketamine in the perioperative period after spine surgery. Loftus et al randomized patients with a history of chronic preoperative opioid use (i.e., daily opiate use for at least 6 weeks) to intraoperative ketamine versus placebo and found a 30% reduction in morphine consumption at 48 hours and an approximately 25% reduction in visual analog scale (VAS) pain score in the post anesthesia care unit and at 6 weeks.4 Although this study provided evidence that there may be reduction in long-term postoperative pain, additional studies are needed to provide evidence that this effect is sustained beyond the 6-week period.

We are interested in examining ketamine more closely in spine surgery because this patient population experiences significant postoperative pain that may be difficult to control due to preoperative opioid use (i.e., opioid tolerance). The investigators chose to study ACDF patients specifically because it is a common spine procedure throughout the United States and the patients have significant opioid requirements postoperatively. In a study examining the effects of the low dose ketamine for postoperative IV PCA fentanyl after cervical and lumbar surgery, patients in the placebo group (and thus only receiving fentanyl PCA) reported mean VAS scores of 4-5 with movement while receiving opioids.5

Further, while previous studies have shown an opioid-sparing effect of ketamine as measured by opioid consumption and a decrease in pain as measured by VAS scores, no study to our knowledge has examined quality of recovery after intraoperative ketamine infusion. The Quality of recovery (QoR-40) score was developed by Myles et al to assess quality of recovery after anesthesia based on forty questions in five dimensions,6 and this score has been shown to be a reliable and valid outcome for patients undergoing both spine and cranial surgery.7 QoR-40 is also of interest because it should be able to provide a global assessment of the possible benefit or harm of using ketamine in patients by simultaneously characterizing the detrimental side effects as well as the positive benefits of ketamine when used as an infusion at subanesthetic levels (studies thus far have shown that there are minimal side effects such as hallucinations).1,4

Significance:

Previous studies have shown an opioid-sparing effect of ketamine, however further research is warranted in patients whose pain may be difficult to control and whether this effect is sustained. ACDF patients experience significant pain post-operatively, and ketamine may improve their quality of recovery due to its opioid-sparing effects and prevention of chronic pain. Further, patient centered outcomes as measured by the QoR-40 have not been reported in the literature when ketamine, or other opioid sparing anesthetics, have been administered. This study will not only determine if the "moderate" dose of ketamine is beneficial or detrimental to the recovery of patients but also whether it can improve long term patient function, presumably by decreasing central pain sensitization. In addition, this study will set the stage for further RCT's examining other analgesic strategies in cervical spine surgery patients (i.e., intraoperative lidocaine infusions, volatile anesthetic vs. propofol as the primary hypnotic, COX-2 inhibitors, pregabalin, etc.). The overall goal would be to develop a multi-faceted regimen that decreases the postoperative inpatient opioid requirements of these patients and may facilitate long term recovery.

The research questions:Does ketamine improve the quality of recovery at 24 hours after anterior cervical discectomy and fusion (ACDF)? The hypothesis: the investigators hypothesize that ketamine will improve the quality of recovery after ACDF surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years)
* Undergoing 1-3 level ACDF surgery

Exclusion Criteria:

* Patients under 18 years of age
* Non-English speaking patients
* Pregnancy
* Emergent procedures
* History of psychosis
* Uncontrolled hypertension
* Known or suspected allergy or intolerance to ketamine or its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery-40 score at 24 hours | 24 hours after surgery
  Quality of recovery survey score completed by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Moreland, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loftus RW, Yeager MP, Clark JA, Brown JR, Abdu WA, Sengupta DK, Beach ML. Intraoperative ketamine reduces perioperative opiate consumption in opiate-dependent patients with chronic back pain undergoing back surgery. Anesthesiology. 2010 Sep;113(3):639-46. doi: 10.1097/ALN.0b013e3181e90914. PMID 20693876